CLINICAL TRIAL: NCT02407522
Title: The Improvements of Dietary Supplement of Black Rice on Metabolic Syndrome and Its Correlation With Metabolism of Gut Microbiota
Brief Title: The Improvements of Dietary Supplement of Black Rice on Metabolic Syndrome
Acronym: IDSBRMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, zhangpeiwen, PhD candidate, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SunYat-senU001
Record Dates: First submitted 2015-03-26; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome; black rice
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- black rice group (Experimental): Each subject in the experimental group will be provided with black rice (50 g/day).According to the clinical requirements, no specific rules are needed for other treatments of the two groups.
  Interventions: Dietary Supplement: Black rice
- white rice group (Placebo Comparator): individuals in the control group will be subjected to follow-up. According to the clinical requirements, no specific rules are needed for other treatments of the two groups.
  Interventions: Other: follow-up

INTERVENTIONS:
Dietary Supplement: Black rice — They asked to keep their normal life style during intervention
  Arms: black rice group
Other: follow-up — They asked not to consume any black rice or excess amount of food rich in anthocyanin compared to their normal life style, such as grapes, blueberry, red wine, black bean during intervention.
  Arms: white rice group

SUMMARY:
The purpose of this study is to thoroughly investigate how the interaction between black rice and human gut microbiota affects metabolic diseases, this study will recruit patients with Metabolic Syndrome (MS) and provide them with dietary supplementation of black rice (50 g/day) for 3 months to observe its effect on the development of MS. The focuses of this project are to elucidate how black rice consumption affects the composition and metabolism of intestinal bacteria as well as the development of MS, and to further analyze whether the changes in intestinal bacteria are associated with the changes in MS improvements.

ELIGIBILITY:
Inclusion Criteria:

* individuals meeting at least 3 of the following 5 criteria will be chosen:
* abdominal obesity: using the waist standard for Asians: waist≥90 for male and ≥80 for female
* high blood sugar: fasting plasma glucose≥5.6mmol/L (100mg/d L) or individuals diagnosed with diabetes and being treated
* hypertension: systolic blood pressure≥130 mm Hg or diastolic blood pressure≥85 mm Hg or individuals diagnosed with hypertension and being treated
* dyslipidemia: fasting total triglycerides≥1.70 mmol/L(150 mg/d L) or individuals undergoing lipid-lowering therapy
* fasting plasma high-density lipoprotein cholesterol<1.03mmol/L (40mg/dL) for male or <1.3mmol/L (50mg/dL) for female.

Exclusion Criteria:

* having current or former cardiovascular disease, including coronary heart disease (e.g., angina pectoris, myocardial infarction, coronary revascularization, abnormal Q waves in ECG), stroke (e.g., congestive, hemorrhagic, or transient ischemic stroke), and intermittent claudication caused by peripheral arterial diseases;
* severe clinical conditions that may compromise patients' participation in experiments, e.g., digestive diseases leading to inability to maintain black rice uptake, patients receiving parenteral nutrition supply, malignancies in progress, and mental illness;
* immunodeficiency disease or AIDS, chronic inflammation conditions
* drug abuse or alcoholism (>80g/d).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
reversal rate of metabolic syndrome | 3 months
  Numerator is number of people is metabolic syndrome at baseline but not after intervention. The denominator is the overall number of people in the group

SECONDARY OUTCOMES:
proportion of Bacteroides | 3months
  PCR analysis the RNA of Bacteroides in faeces
proportion of Bifidobacterium | 3months
  PCR analysis the RNA of Bacteroides in faeces

OTHER OUTCOMES:
changes in fasting blood-glucose | 3 months
  (after intervention - baseline)/baseline×100%
changes in fasting total triglyceride | 3 months
  (after intervention - baseline)/baseline×100%
changes in fasting HDL-c | 3 months
  (after intervention - baseline)/baseline×100%
changes in fasting LDL-c | 3 months
  (after intervention - baseline)/baseline×100%
changes in fasting waistline | 3 months
  (after intervention - baseline)/baseline×100%

CONTACTS AND LOCATIONS:
Overall Officials: Ling wenhua, profess, Study Director — Sun Yat-sen University